CLINICAL TRIAL: NCT07308249
Title: Research on the Application of Brain Network Functional Connectivity Analysis Based on Functional Magnetic Resonance Imaging in Proprioceptive Training for Chronic Non-Specific Low Back Pain
Brief Title: Brain Network fMRI Analysis in Proprioceptive Training for Chronic Low Back Pain
Status: Not yet recruiting | Type: Observational
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: KY-2025-304
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Brain Network Functional Connectivity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Multimodal Imaging Evaluation — Functional connectivity analysis of brain networks based on functional magnetic resonance imaging (fMRI) technology

SUMMARY:
Through longitudinal analysis of dynamic changes in DMN functional connectivity before and after sensory training intervention, combined with pain behavioral and functional improvement indicators, this study systematically reveals the central neural remodeling patterns in CNLBP and establishes an objective efficacy evaluation system based on multimodal imaging.

DETAILED DESCRIPTION:
This phase of the research aims to elucidate the neuroplasticity mechanisms induced by CNLBP treatment, providing a theoretical basis for the future development of personalized rehabilitation protocols based on brain network subtypes, ultimately achieving the clinical goals of reducing pain recurrence rates and improving long-term prognosis in patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years old;

  * Current or past low back pain lasting more than three months; ③ No abnormal sensation or reflex abnormalities in the lower limbs; ④ Able to commit to participating in training three times per week for three months.

Exclusion Criteria:

* Fractures, dislocations, structural abnormalities, prior surgery, metal implants, or lumbar disc herniation;

  * Comorbidities such as severe cardiovascular diseases, neurological disorders, osteoporosis, or metabolic diseases; ③ Low back pain caused by visceral diseases;

    * VAS score (range 1-10) exceeding 8 points;

      * Pregnant or lactating women; ⑥ Symptoms of nerve root irritation; ⑦ Recent participation in core stability training.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All patients were assigned numbers from 1 to 40. Starting at any row and column in a random number table, 40 random numbers were sequentially recorded in correspondence with the patient numbers. The random numbers were then ranked in ascending order, with ranks 1-20 assigned to the experimental group and ranks 21-40 to the control group. All patients continued to receive conventional treatment and comprehensive rehabilitation therapy.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
VAS | After 4 weeks of treatment
  The Visual Analogue Scale (VAS) was used to assess the severity of low back pain, with 0 indicating no pain and 10 indicating unbearable severe pain.
JOA | After 4 weeks of treatment
  The Japanese Orthopaedic Association (JOA) efficacy assessment criteria for low back disorders were applied to evaluate lumbar function.

SECONDARY OUTCOMES:
MRI | After 4 weeks of treatment
  Magnetic resonance imaging was used to assess the effects of treatment on brain networks.

IPD SHARING:
Plan to Share IPD: Undecided